CLINICAL TRIAL: NCT01546558
Title: A Phase 1, Open-label, Single Cohort, Two-Period Fixed Sequence Study to Assess the Pharmacokinetics of Metformin Alone and in Combination With Ranolazine 500 mg Twice Daily in Subjects With Type 2 Diabetes Mellitus
Brief Title: Single Cohort, 2-Period Study to Assess Pharmacokinetics of Metformin Alone and in Combination With Ranolazine 500 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: GS-US-259-0143
Record Dates: First submitted 2012-02-27; First posted 2012-03-07 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Metformin; Ranolazine; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Ranolazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin, Ranolazine (Experimental): Single cohort, 2-period study:
  * Period 1, metformin 1000 mg bid on Days 1-5
  * Period 2, metformin 1000 mg bid + ranolazine 500 mg bid on Days 6-10
  Interventions: Drug: Metformin; Drug: Ranolazine

INTERVENTIONS:
Drug: Metformin — Metformin 1000 mg bid on Days 1-10
  Other Names: Glucophage
Drug: Ranolazine — Ranolazine 500 mg bid on Days 6-10
  Other Names: Ranexa

SUMMARY:
The purpose of this study is to evaluate the effect of steady-state ranolazine 500 mg bid on the steady state pharmacokinetics (PK) of metformin in subjects with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
The primary objective of this study is as follows:

• To evaluate the effect of steady-state ranolazine 500 mg twice daily (bid) on the steady state pharmacokinetics (PK) of metformin in subjects with T2DM.

The secondary objectives of this study are as follows:

* To examine the safety and tolerability of metformin when co administered with ranolazine 500 mg bid at steady-state in subjects with T2DM.
* To determine the steady-state PK of ranolazine 500 mg bid in subjects with T2DM receiving metformin.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 30 to 65 years old, inclusive
* Documented history of T2DM
* HbA1c 6.5%-10%, inclusive
* Fasting serum glucose ≤ 270 mg/dL at Screening
* Fasting C-peptide ≥ 1 ng/mL at Screening
* Stable metformin monotherapy (metformin ≥ 1500 mg total daily dose for at least 4 weeks prior to Screening)
* Body mass index (BMI) 25 to 40 kg/m2, inclusive, at Screening
* Creatinine Clearance > 80 mL/min at Screening
* Females of child-bearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1 and must agree to use highly effective contraception methods from Screening throughout the duration of the Treatment Period and for 14 days following the last dose of study drug

Exclusion Criteria:

* Type 1 Diabetes Mellitus (T1DM)
* Use of insulin therapy < 3 months prior to Screening
* History of ketoacidosis, ketosis-prone diabetes, or lactic acidosis
* Clinically significant complications of diabetes
* History of hypoglycemia
* Any non-insulin antidiabetic therapy (other than metformin) < 2 months prior to Screening
* Any clinically significant cardiovascular event < 2 months prior to Screening
* Clinically significant, inadequately controlled, or unstable hypertension
* Hospitalization < 2 months prior to Screening or major surgery < 3 months prior to Screening
* History of gastrointestinal disease or surgery that could impact drug absorption
* History of substance of alcohol or substance abuse
* Positive urine drug screen for drugs of abuse
* Positive alcohol breath test
* Any other clinically significant existing medical or psychiatric condition or one requiring further evaluation
* Treatment with selected medications
* Hemoglobin < 12 g/dL for males; or < 11 g/dL for females at Screening
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5x upper limits of normal
* Clinically significant history of hepatic disease or evidence of hepatic impairment
* Positive blood screen for hepatitis C or hepatitis B
* QTc interval > 500 msec at Screening
* Females who are pregnant or are breastfeeding

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of metformin | 0, 0.5, 1,1.5, 2, 3, 4, 6, 8, 10 and 12 hours post-dose on Days 5 and 10
Area under the plasma concentration vs time curve over the dosing interval, at steady state (AUCtau) of metformin | 0, 0.5, 1,1.5, 2, 3, 4, 6, 8, 10 and 12 hours post-dose on Days 5 and 10

SECONDARY OUTCOMES:
Number of participants with adverse events | From time of signed informed consent to time of follow-up phone call, an expected average of 5 weeks
Maximum observed plasma concentration (Cmax) of ranolazine and metabolites | 0, 0.5, 1,1.5, 2, 3, 4, 6, 8, 10 and 12 hours post-dose on Day 10
Area under the plasma concentration versus time curve over the dosing interval, at steady state (AUCtau) of ranolazine and metabolites | 0, 0.5, 1,1.5, 2, 3, 4, 6, 8, 10 and 12 hours post-dose on Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Axel Juan, MD, Principal Investigator — SeaView Research, Inc.
Locations (1):
- SeaView Research Inc., Miami, Florida, United States